CLINICAL TRIAL: NCT02188498
Title: Electrocardiography Data Analysis in Sleep Disorders
Acronym: Holter
Status: Completed | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Other Study IDs: Electrocardiography Study
Record Dates: First submitted 2014-07-02; First posted 2014-07-11 (Estimated); Last update posted 2019-01-04 (Actual); Status verified 2019-01

CONDITIONS: Sleep Disorders; Sleep Apnea; Sleep Disordered Breathing
MeSH Terms: conditions — Sleep Wake Disorders; Sleep Apnea Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Polysomnography with Holter monitoring: Patients will undergo resting electrocardiogram (ECG) test at the beginning of the night and be monitored by a Holter device for the duration of the sleep study.
  Interventions: Procedure: Polysomnography

INTERVENTIONS:
Procedure: Polysomnography — Polysomnography, also called a sleep study, is a test used to diagnose sleep disorders. Polysomnography records your brain waves, the oxygen level in your blood, heart rate and breathing, as well as eye and leg movements during the study.

SUMMARY:
The objective of this study is to determine if a non-invasive technique, using an innovative analysis of electrocardiogram (ECG) data, would allow for detection of respiratory events during sleep and discrimination between central and obstructive apnea. Obstructive Sleep Apnea (OSA) is the most common respiratory disturbance seen during sleep, with an estimated prevalence of 10 % in the population and is strongly associated with the development of cardiovascular disease. In patients with underlying cardiac disease, particularly in heart failure (HF), central respiratory events such as Cheyne-Stokes Respiration (CSR) are often seen during sleep. The presence of CSR is also associated with increased cardiovascular morbidity and mortality. Currently, the identification and classification of sleep related respiratory disturbances is performed during over-night sleep studies (polysomnography), which are labor-intensive, time-consuming, expensive and difficult for patients. Thus, the development of alternative techniques to assist in the identification of those events in the outpatient setting is of marked importance for widespread screening of sleep apnea.

DETAILED DESCRIPTION:
This study aims to use novel analyses of electrocardiogram data to detect the presence and type of respiratory event observed in patients during sleep. Our specific aims include: determining the accuracy of using a non-invasive electrocardiogram (ECG) to detect sleep apnea and to distinguish between obstructive sleep apnea (OSA) and Cheyne-Stokes Respiration (CSR). For this investigator-initiated study, data from approximately 400 consecutive patients presenting to the Weill Cornell Center for Sleep Medicine for polysomnography will be collected. A sample size of 45 subjects in each group will be needed to quantify mean amplitude change in the ECG derived respiratory signal. Study procedures are outlined below. Standard and novel, research measurements from the ECG will be correlated with findings from polysomnography and used to assess the presence and severity of a variety of ECG-based measures of cardiovascular disease, such as left ventricular hypertrophy and prior Q-wave myocardial infarction. Subjects will also have to complete a Questionnaire prior to their ECG at their visit.

Detailed procedures:

1. Subjects will be asked to complete a brief questionnaire (see attached). This questionnaire will ask questions relating to subjects' sleep patterns, etc. Potential risks include possible discomfort while completing the questionnaire.
2. Continuous 12-lead ECG recordings, using torso-located electrodes, will be obtained with Mortara Instrument H12+ recorders. An MTA Agreement has been established for the use of this equipment for the duration of this study. Electrocardiograms will be obtained in standard clinical fashion using GE Medical Systems equipment. Patients will be asked to lie in the supine position and 10 recording electrodes will be applied. With the patient lying quietly, a 10 second digital ECG will be recorded and then downloaded via analog modem to the MUSE ECG analysis and storage system at New York Presbyterian Hospital where it will be stored on a dedicated site of our password protected MUSE server. ECG information:12-lead ECGs will be downloaded from the MUSE system to a secure network drive and then copied to the hard drive of a password protected computer where they will be batch-analyzed using an ECG research analysis program, Magellan, provided by GE Medical Systems. Magellan will generate a series of measurements from each ECG and will then export these measurements to an Excel file which will be converted to SPSS files for data analysis. Deidentified ECG data may be downloaded to the Electrocardiography data center and transferred using a secure file transfer system, such as Cornell's file transfer website, to an outside company (Mortara, Inc.) for further analysis as needed.
3. Standard polysomnography will be performed for 12 hours at approximately the patients regular sleep time. Sleep data will be recorded in a digitized system and analyzed using Grass Twin software ® (Middleton, WI) for the determination and classification of respiratory events and other sleep related parameters. The Apnea-Hypopnea Index (AHI) will be calculated by computing the average number of obstructive apneas plus obstructive hypopneas per hour of sleep. Obstructive sleep apnea (OSA) is here defined by an AHI ≥5. Intermittent hypoxemia (IH) will be determined by the number of periods ≥6 sec with SaO2 drops ≥4%. Cheyne-Stokes Respiration will be determined by the typical crescendo-decrescendo pattern on the respiratory flow signal, chest and thoracic impedance, using standard criteria. Total duration of CSR will be calculated for the determination of the % of sleep time on CSR. Data regarding percentage of sleep time at SaO2 ≤90% (%TST<90) and lowest saturation level (LowSaO2) will also be recorded.

Upon completion of data attainment some de-identified data will be remote analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting to the WCMC Sleep Center for polysomnography

Exclusion Criteria:

* N/A

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients undergoing overnight sleep studies
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2013-09; Primary Completion 2017-11 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Heart rate variability | One night of sleep study
  The variation in the time interval between heartbeats. It is measured by the variation in the beat-to-beat interval.

SECONDARY OUTCOMES:
Analysis of QRS morphology | One night of sleep study
  The variation in the QRS waves.
electrocardiogram signal | One night of sleep study
  Variation and analysis in the ecg signal.

CONTACTS AND LOCATIONS:
Overall Officials: Ana Krieger, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Center for Sleep Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No